CLINICAL TRIAL: NCT01483066
Title: A Prospective, Randomized, Post-market, Multi-center Study and Cost-effectiveness Analysis of ShapeMatch Technology A Prospective, Randomized, Post-market, Multi-center Study and Cost-effectiveness Analysis of ShapeMatch Technology
Brief Title: Clinical Outcomes and Cost-effectiveness Analysis of ShapeMatch Technology
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: FDA recall - Canadian system did voluntary suspension of study; Investigators subsequently decided to terminate the study
Sponsor: University of Alberta (Other)
Collaborators: Stryker Canada LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00024283
Record Dates: First submitted 2011-11-25; First posted 2011-12-01 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ShapeMatch Instrumentation (Experimental)
  Interventions: Device: ShapeMatch Technology
- Usual Instrumentation (Active Comparator)
  Interventions: Device: ShapeMatch Technology

INTERVENTIONS:
Device: ShapeMatch Technology — ShapeMatch Technology places a plastic cutting guide on the end of the femur and tibia, so that cuts that do not automatically default to the mechanical axis, but rather attempt to recreate the patient's anatomic alignment.

SUMMARY:
The currently held belief is that total knee replacement (TKR) requires the restoration of the overall limb alignment to coincide with the mechanical limb axis. To align the knee implants with this mechanical axis, rods are used to orient cutting guides with the mechanical axis as defined by the center of the femoral head and talus. Standard surgical technique typically involves femoral and tibial rods with cutting blocks to facilitate the intraoperative alignment of the initial femoral and tibia bone cuts. This approach is the method used for the traditional TriathlonÒ instrumentation. The Patient Specific Cutting Guides are designed to offer an alternative for alignment rods. ShapeMatch Technology places a plastic cutting guide on the end of the femur and tibia, so that cuts that do not automatically default to the mechanical axis, but rather attempt to recreate the patient's anatomic alignment. The surgeon can then assess implant placement and adjust as necessary during pre-operative planning. Thus, Patient Specific Cutting Guides give the surgeon better control over the placement of the implants.

This study will be a prospective, randomized evaluation of ShapeMatch Technology for primary TKR in a consecutive series of patients who meet the eligibility criteria. The clinical study will be accompanied by a formal cost-effectiveness analysis of one-year outcomes.

One half of the cases enrolled will receive the Triathlon® Cruciate Retaining Total Knee System (Triathlon® CR) in a procedure using patient-specific cutting guides designed to reproduce the natural kinematic alignment of the knee. The other half of the cases will receive the Triathlon® CR device in a procedure using traditional instrumentation, without navigation, designed to produce a neutral mechanical alignment. Subjects will be evaluated using validated measures within 3 months prior to surgery and at 6 weeks, 3 months, and 1 and 2 years postoperatively.

Primary Hypothesis:

The investigators expect that ShapeMatch Technology will be as cost-effective as usual care.

Secondary Hypotheses:

The investigators expect that ShapeMatch Technology will result in improved clinical outcomes relative to usual care at three months postoperatively.

The investigators expect that ShapeMatch Technology will result in similar clinical outcomes relative to usual care at two-years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a male or non-pregnant female age 18 to 80 years of age at the time of study device implantation.
* Patient has primary diagnosis of Non-Inflammatory Degenerative Joint Disease (NIDJD).
* Patient is a candidate for a primary total knee replacement (TKR).
* Patient is willing and able to comply with preoperative Magnetic Resonance Imaging (MRI) requirements, postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

* Patient has a Body Mass Index (BMI) ≥ 40.
* Patient has a varus or valgus deformity greater than 10 degrees or flexion contracture greater than 20o.
* Patient has an active or suspected latent infection in or about the affected joint at time of study device implantation.
* Patient has received any orthopaedic surgical intervention to the lower extremities within the past year or is expected to require any orthopaedic surgical intervention to the lower extremities, other than the TKR to be enrolled in this study, within the next year.
* Patient requires bilateral TKR, or has had a contralateral partial TKR or TKR.
* Patient has any implanted device that would be incompatible with MRI procedures.
* Patient has a neuromuscular or neurosensory deficiency, which limits the ability to evaluate the safety and efficacy of the device.
* Patient is diagnosed with a systemic disease (e.g. Lupus Erythematosus) or a metabolic disorder (e.g. Paget's Disease) leading to progressive bone deterioration.
* Patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements(e.g. > 30 days).
* Patient requires revision surgery of a previously implanted total knee replacement or knee fusion to the affected joint.
* Patient has a known sensitivity to device materials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06-26 (Actual); Study Completion 2015-06-26 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness analysis (CEA) | surgery to one year postoperatively
  The CEA will examine the cost of health care resources and health outcomes from the surgical intervention to 1-year postoperatively. The costs will include all health care utilization during this time. Health care utilization, and associated costs, related to the patients' condition, the surgery and adverse events of the surgery will be the basis of a sensitivity analysis.
  Quality adjusted life years (QALYs) is the preferred measure for CEA. QALYs will be calculated based on the EuroQol-5D (EQ-5D). An objective outcome measure may be used for additional analysis.

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | preoperative - 2 years postoperative
  The KOOS is an instrument used to assess the patient's opinion about his or her knee and associated problems and has been validated for use in this population.
EuroQol-5D (EQ-5D) | preoperative to 2-years postoperative
  The EQ-5D is a generic health status questionnaire that will be used to measure overall health status and will be used in the CEA.
University of California at Los Angeles (UCLA) Activity Scale | preoperative to 2-years postoperative
  The UCLA activity score is a self-administered patient evaluation designed to reflect patient activity.
Forgotten Joint Score | Imediate postoperative to 2 years postoperative
  The Forgotten Joint Score is a recently developed tool that examines how aware the subject is of their TKR during activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Arnett, MD, FRCS (C), Principal Investigator — Alberta Health services; Lauren Beaupre, PT, PhD, Study Director — University of Alberta
Locations (1):
- Alberta Health Services - Edmonton zone, Edmonton, Alberta, Canada